CLINICAL TRIAL: NCT04580160
Title: Venous Stent for the Iliofemoral Vein Investigational Clinical Trial Using the DUO Venous Stent System
Acronym: VIVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vesper Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-CA-0001
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: May-Thurner Syndrome; Deep Vein Thrombosis; Chronic Venous Insufficiency
MeSH Terms: conditions — May-Thurner Syndrome; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Duo Venous Stent System Implantation (Experimental)
  Interventions: Device: Duo Venous Stent System

INTERVENTIONS:
Device: Duo Venous Stent System — Subjects with nonmalignant iliofemoral venous outflow obstruction presenting with nonthrombotic (NT), acute thrombotic (AT) or chronic postthrombotic (CPT) disease pathogenesis will be selected for study participation.

SUMMARY:
This is a prospective, multi-center, single-arm, non-blinded clinical trial designed to investigate the safety and efficacy of the Vesper DUO Venous Stent System as compared to a pre-defined performance goal (PG) established from published, peer reviewed scientific literature related to stenting of iliofemoral venous outflow obstructions.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-breastfeeding females ≥18 years of age at the time of consent
2. Subject is able and willing to provide written informed consent prior to receiving any non-standard of care, protocol specific procedures
3. Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to treatment and must use some form of contraception (abstinence is acceptable) throughout the time of clinical trial exit
4. Willing and capable of complying with all required follow-up visits
5. Estimated life expectancy ≥1 year
6. Subject is ambulatory (use of assistive walking device such as a cane or walker is acceptable)
7. Body mass index (BMI) <40
8. Clinically significant symptomatic venous outflow obstruction in one iliofemoral venous segment (one limb) per subject, is indicated for venoplasty and stenting, and meets at least one of the following clinical indicators:

   1. Clinical-Etiology-Anatomy-Pathophysiology (CEAP) score ≥3
   2. Venous Clinical Severity Score (VCSS) pain score ≥2
   3. Suspected deep vein thrombosis (DVT) with symptoms occurring prior to receiving a DUO Stent
9. Subject is willing and able to comply with PI recommendation for compression therapy, if required
10. Presence of unilateral, non-malignant venous obstruction of the common femoral vein (CFV), external iliac vein (EIV), common iliac vein (CIV), or any combination thereof, defined as a ≥50% reduction in target vessel lumen diameter and confirmed by venographic or IVUS imaging. The cranial point of the obstruction may extend to the iliac vein confluence of the inferior vena cava (IVC) and the caudal point may be 2mm above either the inflow of the deep femoral (or profunda) or the lesser trochanter, whichever is most cranial
11. Obstructive lesion(s) able to be treated with continuous stent coverage
12. Adequate inflow to the target lesion(s) involving at least a patent femoral or deep femoral vein and a landing zone in the CFV free from significant disease requiring treatment
13. Reference vessel diameter is of adequate size to accommodate the appropriate size stent as measured by IVUS
14. All vessels from insertion site through target vessel can accommodate a 9F or 10F sheath, depending on the stent size used
15. Ability to cross interventional devices through target lesion(s)
16. In DVT subjects, successful treatment of acute thrombus must have occurred prior to receiving any DUO Stents for an underlying obstructive lesion. Successful treatment of acute thrombus is defined as reestablishment of antegrade flow with ≤30% residual thrombus (confirmed by venogram or IVUS) and freedom from bleeding and symptomatic pulmonary embolism (confirmed by imaging). After successful treatment of thrombus is confirmed, eligible obstructive lesion(s) can be treated with a DUO Stent during the same procedure.
17. All subjects must undergo a SARS-CoV-2 test and have a negative test result within 8 days of the index procedure. If a SARS-CoV-2 test is unavailable due to institution policy, a test shortage, or if there is a delay in test results, the subject must complete the COVID-19 questionnaire and must have answered NO to all questions to be eligible for enrollment. A SARS-CoV-2 test will not be required for enrollment if a subject has received a complete cycle of an authorized COVID-19 vaccine or has documented evidence of a positive COVID-19 antibody test and is asymptomatic and has no long-lasting effects (per PI discretion) from a prior COVID-19 infection.
18. A measured temperature less than 99.5°F (37.5°C) on the day of the index procedure and no history of fever or feeling feverish within 14 days of the index procedure
19. No prior history, within 60 days of the index procedure, of a SARS-CoV-2 positive test, or COVID-19 symptoms

Exclusion Criteria:

1. Target limb symptoms caused by peripheral arterial disease
2. Presence of unresolved significant pulmonary embolism prior to use of the DUO Venous Stent System confirmed by chest CT. If subject has documented history of significant pulmonary embolism within the last 6 months, a chest CT is required to confirm significant pulmonary embolism is not currently present.
3. Presence of IVC obstruction or target venous obstruction that extends into the IVC
4. Presence of acute DVT located outside target limb
5. Contralateral venous occlusive disease of the CFV, EIV, and/or CIV, with planned treatment ≤390 days after the index procedure
6. Uncontrolled or active coagulopathy or known, uncorrectable bleeding diathesis
7. Coagulopathy causing INR >2 which is not amenable to medical treatment
8. Platelet count <50,000 cells/mm3 or >1,000,000 cells/mm3 and/or White blood cell (WBC) <3,000 cells/mm3 or >12,500 cells/mm3
9. Uncorrected hemoglobin of ≤9 g/dL
10. Subject is on dialysis or has an estimated glomerular filtration rate (eGFR) <30 mL/min. In subjects with diabetes mellitus, eGFR <45 mL/min.
11. History of Heparin Induced Thrombocytopenia
12. Presence of known aggressive clotting disorders such as Lupus Anticoagulant Disorder, Antiphospholipid antibody syndrome, homozygous gene Factor V Leiden or Prothrombin gene abnormalities, Protein C and S deficiency or Antithrombin deficiency
13. Known hypersensitivity or contraindication to antiplatelet therapy or anticoagulation, nickel, or titanium
14. Contrast agent allergy that cannot be managed adequately with pre-medication
15. Intended concurrent adjuvant procedure (except for venoplasty) such as creation of temporary arteriovenous fistula, femoral endovenectomy or saphenous vein ablation and/or saphenous vein stripping during the index procedure
16. Subjects who have had any prior surgical or endovascular procedures to the target vessel. Note that subjects who have had successful catheter-directed or mechanical thrombolysis in the target vessel for DVT at least 90 days prior to the index procedure may be included
17. Planned surgical or interventional procedures of the target limb (except thrombolysis and/or thrombectomy in preparation for the procedure or vena cava filter placement prior to stent implantation in subjects at high risk for pulmonary embolism) within 30 days prior to or 30 days after the index procedure
18. Planned surgical or interventional procedures for other medical conditions (i.e., not associated with the target limb) 30 days prior to or 30 days after the index procedure
19. Previous venous stenting of the target limb, the IVC, or contralateral limb if stents extend into the IVC
20. Iliofemoral venous segment unsuitable for treatment with available sizes of DUO Stent implants
21. Lesions with intended treatment lengths extending into the IVC
22. No safe landing zone at or above the profunda femoral confluence
23. Participating in another investigational study in which the subject has not completed the primary endpoint(s)
24. Has other comorbidities that, in the opinion of the Investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2025-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (28):
  - St. Joseph Hospital, Orange, California
  - Stanford University, Palo Alto, California
  - The Vascular Experts, Darien, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center of Florida, Miami, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - University Clinical Research-Deland LLC, Winter Park, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Cardiovascular Institute of the South, Opelousas, Louisiana
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - Edgewood Hospital and Medical Center, Englewood, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Atrium Health, Charlotte, North Carolina
  - The Ohio Health Research Institute, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Houston Healthcare Medical Center, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Hurricane Cardiology Research, New Braunfels, Texas
  - Sentara Clinical Research, Norfolk, Virginia
  - Lake Washington Vascular, PPLC, Bellevue, Washington
  - Medical College of Wisconsin, Vascular & Interventional Radiology, Froedtert Hospital Radiology, Rm 2803, Milwaukee, Wisconsin
- Poland (2):
  - University Hospital in Opole, Opole
  - Medical University of Karol Marcinkowski, Poznan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Duo Venous Stent System: Use of the Duo Venous Stent System in the iliofemoral veins for the treatment of symptomatic venous outflow obstruction.
Period: Overall Study
Arm/Group | Duo Venous Stent System
Started | 162 (Intent to Treat (ITT) population)
Completed | 136 (Completed 12-month follow-up)
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Duo Venous Stent System
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 134
  More than one race | 0
  Unknown or Not Reported | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.7)
CEAP Clinical Assessment [Count of Participants; unit: Participants] — The CEAP (Clinical, Etiological, Anatomical, and Pathophysiological) classification system allows universally uniform diagnosis and comparison of chronic venous disorders. The Clinical aspect of the CEAP classification was used to categorize venous disease. The 'Clinical' signs of venous disease are those that are visible and used to categorize the subject from C0 (No visible or palpable signs of venous disease) to C6r (Recurrent active venous ulcer).
  Participants
    C0 (No visible or palpable signs of venous disease) | 2
    C1 (Telangiectasia or reticular veins) | 1
    C2 (Varicose veins) | 1
    C2r (Recurrent varicose veins) | 0
    C3 (Edema) | 107
    C4 (Changes in skin and subcutaneous tissue secondary to chronic venous disease) | 9
    C4a (Pigmentation or eczema) | 21
    C4b (Lipodermatosclerosis or atrophie blanche) | 3
    C4c (Corona phlebectatica) | 0
    C5 (Healed) | 8
    C6 (Active venous ulcer) | 9
    C6r (Recurrent active venous ulcer) | 1
VCSS Pain [Count of Participants; unit: Participants] — The Venous Clinical Severity Score (VCSS) system is a scoring system used to categorize nine attributes of venous disease. For this study, only the Pain Score was collected. The levels of pain severity ranged from 0 (none) to 3 (severe). Population: VCSS Pain Score is missing for two subjects.
  Participants
    number analyzed (Participants) | 160
    0 - none | 11
    1 - mild (occasional, not restricting activity or requiring analgesics) | 24
    2 - moderate (daily, moderate activity limitation, occasional analgesics) | 84
    3 - severe (daily, severe limiting activities or requiring regular use of analgesics) | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants Free From Major Adverse Events (MAEs) at 30 Days
Description: Freedom from major adverse events (MAEs) at 30 days post index procedure, as adjudicated by the Clinical Events Committee (CEC) or Core Laboratory, including:
  * Device or procedure-related death
  * Device or procedure-related bleed at the target vessel and/or the target lesion or at the access site requiring surgical or endovascular intervention or blood transfusion of ≥2 units
  * Device or procedure-related venous injury occurring in the target vessel and/or the target lesion or at the access site requiring surgical or endovascular intervention
  * Major amputation of the target limb
  * Clinically significant pulmonary embolism (PE), confirmed by CT angiography
  * Stent embolization outside of the target vessel
  * Presence of new thrombus within the stented segment requiring surgical or endovascular intervention
Time Frame: 30 days
Population: The number of evaluable subjects for the 30 day Primacy Safety Endpoint was 159.
Measure: Count of Participants; unit: Participants
Arm/Group | Duo Venous Stent System
Number analyzed (Participants) | 159
Participants | 157

2. Primary Outcome: Efficacy - Number of Participants With Primary Patency of Stented Segment at 12 Months
Description: Primary patency of stented segment at 12 months defined as freedom from:
  * Duplex Ultrasound (DUS) core laboratory adjudicated occlusion or stenosis >50% within the stented segment. If DUS shows >50% stenosis or occlusion, confirmation by diagnostic intravascular ultrasound (IVUS) is required.
  * CEC adjudicated clinically driven target lesion reintervention (CD-TLR) defined as endovascular or surgical procedure for new, recurrent, or worsening symptoms and core lab adjudicated >50% stenosis or occlusion within the stented segment confirmed by diagnostic IVUS
Time Frame: 12 months
Population: Of the 136 subjects that completed 12-month follow-up, 132 had data evaluable for the 12-month primary efficacy endpoint. The four subjects in question did not complete the 12-month DUS or had a non-diagnostic 12-month DUS.
Measure: Count of Participants; unit: Participants
Arm/Group | Duo Venous Stent System
Number analyzed (Participants) | 132
Participants | 119

3. Secondary Outcome: VCSS Pain Score and Changes in VCSS From Baseline in ITT Patients
Description: The Venous Clinical Severity Score (VCSS) system is a scoring system used to categorize nine attributes of venous disease. For this study, only the Pain Score was collected. The levels of pain severity ranged from 0 (none) to 3 (severe).
Time Frame: 12 months
Population: Although 136 subjects completed 12-month follow-up, two additional subjects completed 12-month telephone visits during which VCSS data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Duo Venous Stent System: Baseline VCSS Pain Score
- DUO Venous Stent System: VCSS Pain Score at 12 months
Arm/Group | Duo Venous Stent System | DUO Venous Stent System
Number analyzed (Participants) | 160 | 138
score on a scale | 2.0 (0.8) | 0.5 (0.8)

4. Secondary Outcome: Number of ITT Subjects With Primary Assisted Patency at 12 Months
Description: Primary assisted patency is defined as freedom from DUS core laboratory adjudicated occlusion or stenosis >50% within the stented segment following a reintervention due to a >50% but <100% stenosis. If DUS shows >50% stenosis or occlusion, confirmation by diagnostic IVUS is required.
Time Frame: 12 months
Population: Primary Assisted Patency data is missing for 5/136 subjects that completed 12-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Duo Venous Stent System
Number analyzed (Participants) | 131
Participants | 124

5. Secondary Outcome: Number of ITT Subjects With Secondary Patency at 12 Months
Description: Secondary patency at 12 months defined as freedom from DUS core laboratory adjudicated occlusion or stenosis >50% within the stented segment following a reintervention due to 100% occlusion. If DUS shows >50% stenosis or occlusion, confirmation by diagnostic IVUS is required.
Time Frame: 12 months
Population: Secondary Patency data is missing for 5/136 subjects that completed 12-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Duo Venous Stent System
Number analyzed (Participants) | 131
Participants | 125

ADVERSE EVENTS:
Time Frame: Summary of adverse events that have been reported through 390 days
Arm/Group | Duo Venous Stent System
All-Cause Mortality (participants affected / at risk) | 2/162
Serious Adverse Events (participants affected / at risk) | 46/162
Other Adverse Events (participants affected / at risk) | 102/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duo Venous Stent System (N=162)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Cardiac Disorders (Cardiac disorders) | 5 (6)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (5)
General disorders and administration site conditions (General disorders) | 7 (7)
Infections and infestations (Infections and infestations) | 8 (9)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (2)
Nervous system disorders (Nervous system disorders) | 3 (5)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Product issues (Product Issues) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 2 (3)
Vascular disorders (Vascular disorders) | 9 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duo Venous Stent System (N=162)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 (6)
Cardiac disorders (Cardiac disorders) | 12 (17)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 2 (3)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 19 (22)
General disorders and administration site conditions (General disorders) | 31 (44)
Immune system disorders (Immune system disorders) | 2 (2)
Infections and infestations (Infections and infestations) | 39 (51)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 13 (14)
Investigations (Investigations) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 32 (47)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Nervous system disorders (Nervous system disorders) | 16 (23)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Product issues (Product Issues) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 4 (5)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 10 (14)
Surgical and medical procedures (Surgical and medical procedures) | 3 (4)
Vascular disorders (Vascular disorders) | 27 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04580160/Prot_SAP_000.pdf